CLINICAL TRIAL: NCT00188968
Title: A Randomized, Controlled Trial of Synchronized Nasal Intermittent Positive Pressure Ventilation Versus Nasal Continuous Positive Airway Pressure Using the Infant Flow Advance to Facilitate Successful Extubation in Premature Infants.
Brief Title: Randomized Trial of Nasal Continuous Positive Airway Pressure or Synchronized Nasal Ventilation in Premature Infants.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Manitoba (Other)
Collaborators: Health Sciences Centre Foundation, Manitoba (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B2004:172
Record Dates: First submitted 2005-09-13; First posted 2005-09-16 (Estimated); Last update posted 2007-05-02 (Estimated); Status verified 2007-04

CONDITIONS: Apnea; Infant, Premature; Bronchopulmonary Dysplasia
Keywords: Xanthines; Reintubation; Nasal Intermittent Ventilation; Nasal continous positive airway pressure
MeSH Terms: conditions — Apnea; Premature Birth; Bronchopulmonary Dysplasia | interventions — Continuous Positive Airway Pressure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: Nasal Continuous Positive Airway Pressure
Procedure: Synchronized Nasal Positive Pressure Ventilation

SUMMARY:
Very premature infants uniformly do not have mature functioning lungs to breathe well nor mature regulation mechanisms to breathe regularly. Assistance with a mechanical respirator is common. However, prolonged use of a respirator can itself cause long-term complications. Furthermore, commonly used drugs to improve the regularity of breathing may have long-term consequence only recently recognized. This study will compare two different types of assistance using a nasally applied breathing assist device. The aim is to see which type of assistance is best at avoiding the need for both prolonged respirator use and drugs to regulate breathing.

DETAILED DESCRIPTION:
Early extubation of premature infants may limit the deleterious effects of positive pressure ventilation. The primary cause of failure of extubation (and the need for reintubation) is apnea of prematurity. Standard treatment for improving extubation success and decreasing apnea of prematurity is with the use of nasal continuous positive airway pressure (nCPAP), use of methylxanthines, or both. Recent literature suggests that methylxanthines may have significant effect on long-term neurodevelopmental outcome.

This primary objective of this study is to investigate the effect of synchronized nasal intermittent positive pressure ventilation (sNIPPV) combined with standard nasal continuous positive airway pressure (nCPAP) versus standard nCPAP alone, on the need for reintubation and the need of methylxanthine therapy in premature infants. The study period for the primary objective will be the first 7 days immediately after the initial extubation of premature infants with birth weights 500-1250 grams. A secondary objective is to identify any differences in duration of time free of endotracheal intubation and duration of time free of methylxanthine use between the two treatment modalities as measured from the first extubation attempt.

The study is a randomized, controlled trial using a new CPAP machine (Infant Flow advance™) that will be able to provide nCPAP with and without sNIPPV. Because of the mechanics of the sNIPPV mode, blinding of the study is not possible. The study is pragmatic in design allowing the medical staff to make clinical decisions on ventilatory management based on the routinely used criteria thus evaluating the study interventions in the everyday clinical environment. Analysis will be on an intention-to-treat basis.

ELIGIBILITY:
Inclusion Criteria:

* Premature infants with birth weight 500-1250 grams
* first attempt at extubation

Exclusion Criteria:(clinical suspicion or documented diagnosis of:

* neuromuscular disease
* chromosomal abnormality
* or any congenital anomalies that would affect ability to be extubated from mechanical ventilation via endotracheal tube (i.e. congenital cardiac anomalies, choanal atresia).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2004-11; Study Completion 2007-02 (Actual)

PRIMARY OUTCOMES:
Need for methylxanthine treatment OR the need for re-intubation in the first 7 days after the initial extubation in preterm infants intubated for treatment of respiratory distress. | 7 days immediately after first extubation attempt

SECONDARY OUTCOMES:
Duration of time to methylxanthine treatment. | During first 7 days and during hospitalization
Duration of supplemental oxygen use | During hospitalization
Incidence of bronchopulmonary dysplasia (both 28 days of age, and 36 weeks PCA) | 28 days of age, 36 weeks PCA
Frequency of apneas during the initial 7 days post-extubation. | Initial 7 days post-extubation
Complications of therapy (air leak syndromes, gastric and intestinal distension). | During Hospitalization

CONTACTS AND LOCATIONS:
Overall Officials: Aaron Chiu, MD, Principal Investigator — University of Manitoba; Ruben Alvaro, MD, Principal Investigator — University of Mantioba
Locations (2):
- Canada (2):
  - Health Sciences Centre, Winnipeg, Manitoba
  - St. Boniface General Hospital, Winnipeg, Manitoba